CLINICAL TRIAL: NCT06964503
Title: Impact of Psychological Stress on Treatment Response and Prognosis in Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, PHD, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: LUNG-MOOD-001
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cancer of Lung; Depression Disorders; Anxiety Disorder/Anxiety State
MeSH Terms: conditions — Lung Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Advanced Stage Cohort
  Interventions: Other: Exposure: psychological stress status
- Early-Stage Surgical Cohort
  Interventions: Other: Exposure: psychological stress status
- neoadjuvant therapy Cohort
  Interventions: Other: Exposure: psychological stress status

INTERVENTIONS:
Other: Exposure: psychological stress status — The assessment of depressive and anxiety symptoms was conducted using Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder Assessment 7 (GAD-7). Patients with a PHQ-9 score ≥ 5 or a GAD-7 score ≥ 5 were categorized as the stressed group.

SUMMARY:
This study explores how psychological stress may influence the treatment response and long-term outcomes in patients with lung cancer. While advances in surgery, chemotherapy, immunotherapy, and targeted therapies have improved survival, emotional well-being remains an often-overlooked factor. We aim to investigate whether high levels of stress, anxiety, or depression at the time of diagnosis or during treatment are linked to poorer responses to therapy or shorter survival. By identifying these associations, the study hopes to highlight the importance of psychological care as part of comprehensive cancer treatment. The findings may inform future strategies to integrate mental health support into routine care for patients with both early-stage and advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria (Advanced Stage Cohort):

Age ≥ 18 years; Histologically confirmed diagnosis of lung cancer (including both non-small cell lung cancer [NSCLC] and small cell lung cancer [SCLC]); Unresectable, locally advanced, metastatic, or recurrent disease classified as stage IIIB-IV according to the 8th edition of the AJCC TNM staging system; Eastern Cooperative Oncology Group (ECOG) performance status of 0-1; No prior systemic treatment (e.g., chemotherapy, anti-angiogenic therapy, targeted therapy, or immunotherapy); At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1); Able to provide informed consent and voluntarily agree to participate in the study.

Exclusion Criteria:

Combined with other malignant tumors in the past 3 years; Concurrent acute or chronic psychiatric disorders; Current receiving anti-depressive or anti-anxiety therapy; Previous treatment with other clinical drug trials; Patients with symptomatic brain metastasis; Can't cooperate with psychological scale assessment;

Inclusion Criteria (Early-Stage Surgical Cohort) Age ≥18 years; Pathologically diagnosed as non-small-cell lung cancer； Pathologically stage conformed as early stage of IA-IIIA Available for tumor tissue samples； Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy ); Receiving radical surgery; Informed and agreed to participate in the study;

Exclusion Criteria:

Combined with other malignant tumors in the past 3 years; Concurrent acute or chronic psychiatric disorders; Current receiving anti-depressive or anti-anxiety therapy; Previous treatment with other clinical drug trials; Can't cooperate with psychological scale assessment;

Inclusion Criteria (neoadjuvant therapy Cohort) Adults aged ≥18 years; Histologically confirmed diagnosis of non-small cell lung cancer [NSCLC]; Clinical stage IB-IIIB based on the 8th edition of the AJCC TNM staging system and deemed potentially resectable after neoadjuvant therapy; At least one measurable lesion can be evaluated according to the RECIST 1.1 standard; Planned to receive or currently receiving neoadjuvant systemic therapy (e.g., chemotherapy, targeted therapy, or immunotherapy) with curative intent; Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 prior to neoadjuvant treatment; No prior systemic treatment before the initiation of neoadjuvant therapy; Able to provide informed consent and voluntarily agree to participate in the study

Exclusion Criteria:

Combined with other malignant tumors in the past 3 years; Concurrent acute or chronic psychiatric disorders; Current receiving anti-depressive or anti-anxiety therapy; Previous treatment with other clinical drug trials; Can't cooperate with psychological scale assessment;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants including the patients diagnosed with advanced non-small-cell lung cancer (NSCLC) who received the first-line therapy or neoadjuvant therapy of ICIs; patients diagnosed with advanced small-cell lung cancer (SCLC) receiving the first-line therapy ICIs; patients diagnosed with early small-cell lung cancer (SCLC) receiving surgery.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2030-05-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Advanced Stage Cohort: Progression-free survival (PFS) | 3 years
  Time from the beginning of first-line immunotherapy to the first progression (PD) in patients with lung cancer
Early-Stage Surgical Cohort: Disease-free survival (DFS) | 5 years
  The duration between the date after surgery to the date of any recurrence or death firstly
neoadjuvant therapy Cohort: Pathologic complete response (pCR) rate | 3 years
  pCR is no viable tumor cells in tumor bed and lymph nodes. The pCR rate is the proportion of patients with a pathologic complete response.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Overall survival (OS) is defined as the duration from the beginning of first-line immunotherapy until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Objective Response Rate (ORR) | 3 years
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

OTHER OUTCOMES:
The correlation between gut microbiota and chronic stress | 5 years
  The baseline faeces is collected and assessed by 16S rRNA sequencing. And explore the association between gut microbiota and chronic stress during the enrolled observation process
The correlation between peripheral stress biomarker and immune cells signature and chronic stress | 5 years
  The baseline peripheral venous blood is collected. The stress biomarkers including epinephrine, cytokines, norepinephrine, cortisol and ACTH. The peripheral immune cells signature and assessed by flow cytometry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and DC cells.
The correlation between tumor microenvironment signature and chronic stress | 5 years
  The baseline paraffin-embedded tissue is collected and assessed by multiplex immunohistochemistry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and DC cells. And explore the association between tumor microenvironment signature and chronic stress during the enrolled observation process.